CLINICAL TRIAL: NCT02675777
Title: Sustained Implementation of Patient-Centered Care for Alcohol Misuse
Brief Title: Sustaining Patient-centered Alcohol-related Care
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AHRQ-R18-HS023173
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Alcohol, Drinking; Alcohol Use Disorder
Keywords: Alcohol misuse; Unhealthy alcohol use; Alcoholism; Alcohol dependence; Alcohol abuse; Risky drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quality Improvement Intervention (Experimental): Quality improvement intervention: 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs (see "Intervention") as part of behavioral health integration.
  Interventions: Other: Quality Improvement Intervention
- Usual Care (No Intervention): Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).

INTERVENTIONS:
Other: Quality Improvement Intervention — Group Health clinical leaders and clinicians implement all aspects of behavioral health integration (screening, assessment, and shared decision-making followed by treatment). The implementation strategy, which was refined during the pilot phase, will include:
  1. Identification of a clinical champion and Local Implementation Team.
  2. Participatory Design.
  3. Training primary care providers and Medical Assistants.
  4. EHR clinical decision support tools
  5. Weekly facilitated Local Implementation Team meetings.
  6. Performance monitoring with feedback, including monthly PDCA meetings with the Local Implementation Team and clinic leaders.
  7. Learning sessions for primary care providers during implementation.
  8. Social worker use of an EHR registry with weekly supervision.
  9. Video and handout explicitly designed to shift attitudes about unhealthy alcohol use (overcoming misconceptions and stigma)
  Arms: Quality Improvement Intervention

SUMMARY:
Alcohol use is the third greatest cause of disability and death for US adults. Care for unhealthy alcohol use is lacking in most primary care settings. This project will implement two types of evidence-based care for unhealthy alcohol use in the 25 primary clinics of a regional health system-Group Health (GH). These include preventive care and treatment. Preventive care consists of alcohol screening, and for patients who screen positive, brief patient-centered counseling. Treatment for alcohol use disorders includes offering shared decision making and motivational counseling designed to enhance engagement in one or more treatment options: counseling, medications, and/or specialty treatment. During a pilot phase, the research team at Group Health Research Institute partnered with Group Health leaders and front line clinicians to design, pilot test, and iteratively refine an implementation strategy in 3 Group Health primary care clinics.

Objective

This study uses state-of-the-art implementation strategies to integrate evidence-based alcohol-related care into 22 primary care clinics (detailed below). This study is a pragmatic stepped-wedge quality improvement trial to evaluate its impact on:

1. The proportion of patients who have primary care visits who screen positive for unhealthy alcohol use and have documented annual brief alcohol counseling;
2. The proportion of patients who have primary care visits who have AUDs identified, and a) initiate and b) engage in care for AUDs.

Secondary outcomes will include:

1. The proportion of patients who have primary care visits who have documented annual alcohol screening with the AUDIT-C; and
2. The proportion of patients who have primary care visits who screen positive for severe unhealthy alcohol use and have AUDs assessed and/or diagnosed;

DETAILED DESCRIPTION:
Group Health's Behavioral Health Service leaders decided to implement alcohol-related care along with integration of population-based primary care for other behavioral health conditions, including screening for depression, marijuana and other substance use and use disorders. Group Health leaders also decided to transition primary care social workers to become integrated behavioral health clinicians in 2015.

Pilot testing of the implementation strategies in 2015 was led by Group Health's Behavioral Health Service (BHS) in collaboration with other Group Health departments. State-of-the-art implementation methods were used to integrate evidence-based alcohol-related care into 3 pilot primary care clinics in Group Health. The implementation strategies included: participatory design, clinical champions, practice facilitation, performance monitoring and feedback, and clinical decision support in the electronic health record (EHR). The implementation strategies also included a video and handout designed explicitly to shift staff attitudes, in order to make discussions of unhealthy alcohol use routine and less stigmatized in primary care. Screening and follow-up assessment for symptoms of AUDs are conducted on paper and then typically entered into the EPIC EHR by medical assistants (MAs). The implementation strategy was refined based on ongoing formative evaluation.

Group Health leaders are now prepared to roll out behavioral health integration to the remaining 22 primary care clinics. All implementation will be led and conducted by Group Health clinical leaders and clinicians. The timing of implementation at the 22 clinics is staggered to allow for support from practice facilitators. Leaders randomized clinics to different start dates to allow a rigorous evaluation using secondary quality improvement data.

The research team at Group Health Research Institute is supporting implementation and will lead the evaluation. The research team will conduct a pragmatic stepped-wedge quality improvement trial in the 22 primary care clinics. Implementation will be staggered in 7 waves, each of which will be 4 months long (3 waves in Year 1; 4 waves in Years 2-3). Randomization is stratified by study Year, with 9 sites chosen by Group Health clinical leaders to start in Year 1, and the 13 remaining sites to be randomized in Year 2. Randomization is stratified primarily because Group Health clinical leaders wanted to choose the first 9 clinics. In addition, they may decide remove 3 or 4 facilities in Spokane (a long distance from Seattle requiring air travel) from the Year 2 randomization (thereby omitting 1 of the 7 waves of implementation Year 2).

Due to the pragmatic nature of this trial, clinical partners requested some modifications to the trial design. Please see the study pilot results, protocol paper, and main results paper for details. Of note, the 22 practices were randomized as 19 "sites" because clinical leaders requested that three pairs of nearby practices be randomized together as 3 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Group Health group practice patients, AND
2. Age 18 years and older, AND
3. Have one or more visits at one or more of the randomized Group Health primary care clinics between February 1, 2016 and August 31, 2018.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Bradley, MD, MPH, Principal Investigator — Group Health Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glass JE, Bobb JF, Lee AK, Richards JE, Lapham GT, Ludman E, Achtmeyer C, Caldeiro RM, Parrish R, Williams EC, Lozano P, Bradley KA. Study protocol: a cluster-randomized trial implementing Sustained Patient-centered Alcohol-related Care (SPARC trial). Implement Sci. 2018 Aug 6;13(1):108. doi: 10.1186/s13012-018-0795-9. PMID 30081930
- [Background] Bobb JF, Lee AK, Lapham GT, Oliver M, Ludman E, Achtmeyer C, Parrish R, Caldeiro RM, Lozano P, Richards JE, Bradley KA. Evaluation of a Pilot Implementation to Integrate Alcohol-Related Care within Primary Care. Int J Environ Res Public Health. 2017 Sep 8;14(9):1030. doi: 10.3390/ijerph14091030. PMID 28885557
- [Background] Lee AK, Bobb JF, Richards JE, Achtmeyer CE, Ludman E, Oliver M, Caldeiro RM, Parrish R, Lozano PM, Lapham GT, Williams EC, Glass JE, Bradley KA. Integrating Alcohol-Related Prevention and Treatment Into Primary Care: A Cluster Randomized Implementation Trial. JAMA Intern Med. 2023 Apr 1;183(4):319-328. doi: 10.1001/jamainternmed.2022.7083. PMID 36848119
- [Derived] Angerhofer Richards J, Cruz M, Stewart C, Lee AK, Ryan TC, Ahmedani BK, Simon GE. Effectiveness of Integrating Suicide Care in Primary Care : Secondary Analysis of a Stepped-Wedge, Cluster Randomized Implementation Trial. Ann Intern Med. 2024 Nov;177(11):1471-1481. doi: 10.7326/M24-0024. Epub 2024 Oct 1. PMID 39348695

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this stepped wedge study, 19 sites were randomly assigned to 7 waves, which determined the time period in which they would implement the Quality Improvement Intervention. This study used an open cohort design, in which patients were analyzed during the time periods in which they had visits to a particating site. Therefore, patients could visit the site in one or both periods (i.e., before and/or after the Quality Improvement Intervention began), and also could visit sites in multiple waves.
Units Other Than Participants: sites
Groups:
- Wave 1: These were the sites randomized to implement the intervention in the first wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 2: These were the sites randomized to implement the intervention in the second wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 3: These were the sites randomized to implement the intervention in the third wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 4: These were the sites randomized to implement the intervention in the fourth wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 5: These were the sites randomized to implement the intervention in the fifth wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 6: These were the sites randomized to implement the intervention in the sixth wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
- Wave 7: These were the sites randomized to implement the intervention in the seventh wave.
  The sites within each wave started in Usual Care and then implemented the Quality Improvement Intervention.
  Usual Care:
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
  Quality Improvement Intervention:
  Care received after active implementation begins and before the end of the study in 7/2018. Active implementation is 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs as part of behavioral health integration.
Period: Usual Care
Arm/Group | Wave 1 | Wave 2 | Wave 3 | Wave 4 | Wave 5 | Wave 6 | Wave 7
Started (Given the open cohort design, these are the patients whose first visit to the participating sites within the given wave occurred during the Usual Care period (Period 1).) | 27543; 3 sites | 34989; 3 sites | 39357; 3 sites | 75377; 3 sites | 35287; 3 sites | 41503; 2 sites | 31248; 2 sites
Completed | 27543; 3 sites | 34989; 3 sites | 39357; 3 sites | 75377; 3 sites | 35287; 3 sites | 41503; 2 sites | 31248; 2 sites
Not Completed | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites
Period: Quality Improvement Intervention
Arm/Group | Wave 1 | Wave 2 | Wave 3 | Wave 4 | Wave 5 | Wave 6 | Wave 7
Started (Given the open cohort design, these are only the patients whose first visit to the sites randomized to each wave occurred during the Quality Improvement Intervention (Period 2). This does not include individuals who started in the Usual Care (Period 1) period and had a subsequent visit during the Quality Improvement Intervention period.) | 23888; 3 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 20146; 3 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 17973; 3 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 23917; 3 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 8837; 3 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 6345; 2 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.) | 2226; 2 sites (This is an open-cohort study so different patients were enrolled during Period 1 vs. Period 2.)
Completed | 23888; 3 sites | 20146; 3 sites | 17973; 3 sites | 23917; 3 sites | 8837; 3 sites | 6345; 2 sites | 2226; 2 sites
Not Completed | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites | 0; 0 sites

BASELINE CHARACTERISTICS:
Population: Patients could have a visit in both periods (total number of patients with a visit = 333,596; number of patients with visits in both periods = 150,451).
Groups:
- Quality Improvement (SPARC) Intervention Period: Primary care patients with visits to clinics during months after the clinic was randomly assigned to launch the quality improvement (SPARC) intervention.
- Usual Care Period: Primary care patients with visits to clinics during months before the clinic was randomly assigned to launch the quality improvement (SPARC) intervention.
- Total: Total of all reporting groups
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period | Total
Number analyzed (Participants) | 228258 | 255789 | 484047
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The populations overlap, so we separated by arm.
  years
    SPARC Intervention Period: number analyzed (Participants) | 228258 | 0 | 228258
    SPARC Intervention Period | 50.20 (18.09) |  | NA (NA) — Populations overlapped due to crossover design.
    Usual Care Period: number analyzed (Participants) | 0 | 255789 | 255789
    Usual Care Period |  | 49.30 (18.10) | NA (NA) — Populations overlapped due to crossover design.
Sex/Gender, Customized [Number; unit: participants] — Population: The populations overlap, so we separated by arm.
  participants
    Female - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Female - SPARC | 135426 |  | 135426
    Female - Usual: number analyzed (Participants) | 0 | 255789 | 255789
    Female - Usual |  | 149557 | 149557
    Male - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Male - SPARC | 92830 |  | 92830
    Male - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Male - Usual Care |  | 106231 | 106231
    Unknown - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Unknown - SPARC | 2 |  | 2
    Unknown - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Unknown - Usual Care |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The populations overlap, so we separated by arm.
  Participants
    SPARC Period: number analyzed (Participants) | 228258 | 0 | 228258
    SPARC Period: Hispanic or Latino | 13362 |  | 13362
    SPARC Period: Not Hispanic or Latino | 203201 |  | 203201
    SPARC Period: Unknown or Not Reported | 11695 |  | 11695
    Usual Care Period: number analyzed (Participants) | 0 | 255789 | 255789
    Usual Care Period: Hispanic or Latino |  | 15086 | 15086
    Usual Care Period: Not Hispanic or Latino |  | 230820 | 230820
    Usual Care Period: Unknown or Not Reported |  | 9883 | 9883
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The populations overlap, so we separated by arm.
  Participants
    Asian - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Asian - SPARC | 24866 |  | 24866
    Asian - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Asian - Usual Care |  | 24806 | 24806
    Black or African American - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Black or African American - SPARC | 12525 |  | 12525
    Black or African American - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Black or African American - Usual Care |  | 14679 | 14679
    Hawaiian or Pacific Islander - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Hawaiian or Pacific Islander - SPARC | 2346 |  | 2346
    Hawaiian or Pacific Islander - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Hawaiian or Pacific Islander - Usual Care |  | 2783 | 2783
    Native American or Alaskan Native - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Native American or Alaskan Native - SPARC | 1635 |  | 1635
    Native American or Alaskan Native - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Native American or Alaskan Native - Usual Care |  | 2042 | 2042
    Multiple Race/Other - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Multiple Race/Other - SPARC | 6749 |  | 6749
    Multiple Race/Other - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Multiple Race/Other - Usual Care |  | 7932 | 7932
    Other - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Other - SPARC | 8619 |  | 8619
    Other - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Other - Usual Care |  | 9212 | 9212
    Unknown - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    Unknown - SPARC | 10754 |  | 10754
    Unknown - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    Unknown - Usual Care |  | 9681 | 9681
    White - SPARC: number analyzed (Participants) | 228258 | 0 | 228258
    White - SPARC | 160764 |  | 160764
    White - Usual Care: number analyzed (Participants) | 0 | 255789 | 255789
    White - Usual Care |  | 184654 | 184654

OUTCOME MEASURES:

1. Primary Outcome: Brief Alcohol Counseling Rate
Description: Among patients who have at least one primary care visit, the proportion who screen positive for unhealthy alcohol use (3 or more points for women and 4 or more for men on the AUDIT-C) and have brief alcohol counseling documented in their EHRs in the 14 days after the screen or in the prior year.
Time Frame: Rates of documented brief alcohol counseling within 14 days after a positive alcohol screen will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial.
Measure: Number; unit: participants per 10,000 with visits
Groups:
- Quality Improvement (SPARC) Intervention Period: Primary care patients with visits to clinics during months after the clinic was randomly assigned to launch the quality improvement (SPARC) intervention.
  Quality improvement (SPARC) intervention: 4 months during which a practice facilitator supports the clinic in implementing routine, population-based screening, assessment, treatment, and follow-up for unhealthy alcohol use and AUDs (see "Intervention") as part of behavioral health integration.
  Quality Improvement (SPARC) Intervention: Group Health clinical leaders and clinicians implement all aspects of behavioral health integration (screening, assessment, and shared decision-making followed by treatment). The implementation strategy, which was refined during the pilot phase, will include:
  1. Identification of a clinical champion and Local Implementation Team.
  2. Participatory Design.
  3. Training primary care providers and Medical Assistants.
  4. EHR clinical decision support tools
  5. Weekly facilitated Local Implementation Team meetings.
  6. Performance monitoring with feedback, including monthly PDCA meetings with the Local Implementation Team and clinic leaders.
  7. Learning sessions for primary care providers during implementation.
  8. Social worker use of an EHR registry with weekly supervision.
  9. Video and handout explicitly designed to shift attitudes about unhealthy alcohol use (overcoming misconceptions and stigma)
- Usual Care Period: Primary care patients with visits to clinics during months before the clinic was randomly assigned to launch the quality improvement (SPARC) intervention.
  Care received after 2/2016 but before active implementation begins, which includes passive access to tools in the EHR and 2 months of preparation in each clinic (team building and local pretesting by a local implementation team supported by the external practice facilitator).
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 57 | 11
Statistical Analysis 1: Comparison: Quality Improvement (SPARC) Intervention Period vs Usual Care Period; Test type: Superiority; p < .001, Mixed Models Analysis

2. Primary Outcome: HEDIS Defined Initiation and Engagement in Care for Alcohol Use Disorders
Description: Among patients who have at least one primary care visit, the proportion who are diagnosed with a new AUD and meet criteria for a) "initiation" and b) "engagement" in care for AUDs (as defined by NCQAs HEDIS measures in 2014) based on care documented in their EHRs or via claims for AUD treatment.
Time Frame: Rates of initiation and engagement will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial.
Measure: Number; unit: participants per 10,000 with visits
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 1.4 | 1.8
Statistical Analysis 1: Comparison: Quality Improvement (SPARC) Intervention Period vs Usual Care Period; Test type: Superiority; p = 0.30, Mixed Models Analysis

3. Secondary Outcome: Alcohol Screening Rate
Description: Among patients who have at least one primary care visit, the proportion who have alcohol screening with the AUDIT-C documented in their EHR on the date of the visit or in the prior year.
Time Frame: Assessment rates will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial
Measure: Number; unit: participants per 10,000 with visits
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 8320 | 2080

4. Secondary Outcome: AUD Assessment Rate
Description: Among patients who have at least one primary care visit, the proportion who screen positive for severe unhealthy alcohol use (AUDIT-C 7-12) and have assessment for AUDs, or an AUD diagnosis, documented in their EHR on the date of the visit or in the prior year.
Time Frame: Screening rates will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial.
Measure: Number; unit: participants per 10,000 with visits
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 80.9 | 4.1

5. Other Pre Specified Outcome: Rate of (New) Diagnosis of Alcohol Use Disorders
Description: New AUD diagnosis meant that International Classification of Diseases, Ninth or Tenth Revision (ICD-9/ICD-10) code for an AUD documented at the visit and no AUD diagnosis in prior year.
Time Frame: Rates of AUD diagnosis will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial.
Measure: Number; unit: participants per 10,000 with visits
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 33.8 | 28.8

6. Other Pre Specified Outcome: AUD Treatment Initiation
Description: AUD treatment initiation meant that a new AUD diagnosis was documented at a visit and treatment was documented in a separate visit on the day of diagnosis or within 14 days after the visit (see article text for definition of treatment).
Time Frame: Rates of AUD treatment initiation will be compared before and after "time one" (T1: the start of the 4 months of active implementation) for the pragmatic stepped-wedge trial.
Measure: Number; unit: participants per 10,000 with visits
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
Number analyzed (Participants) | 228258 | 255789
participants per 10,000 with visits | 7.8 | 6.2

7. Other Pre Specified Outcome: Maintenance of Alcohol-related Care
Description: Rates of all primary and secondary outcomes (above) will be compared before and after "time two" (T2: the end of the 4 months of active support for implementation) for the pragmatic stepped-wedge trial.
Time Frame: Rates of all primary and secondary outcomes (above) will be compared before and after "time two" (T2: the end of the 4 months of active support for implementation) for the pragmatic stepped-wedge trial.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: N/A, adverse events were not collected for this pragmatic quality improvement implementation trial. All clinical care was under the purview of the health system.
Description: N/A, adverse events were not collected for this pragmatic quality improvement implementation trial. All clinical care was under the purview of the health system.
Arm/Group | Quality Improvement (SPARC) Intervention Period | Usual Care Period
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT02675777/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT02675777/SAP_001.pdf